CLINICAL TRIAL: NCT01960452
Title: A High Density EEG Comparison of Sleep, Sleep Initiation, and Arousal Patterns in Insomnia Patients and Normal Controls
Brief Title: A High Density EEG Comparison of Sleep Patterns in Insomnia
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-1613; HSC-2013-0019 (Other: UW IRB (Tononi))
Record Dates: First submitted 2013-10-04; First posted 2013-10-10 (Estimated); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Primary Insomnia
Keywords: Insomnia; Primary insomnia; High density EEG; Polysomnography; Healthy sleeping controls
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary insomnia: Participants classified as having insomnia through clinical interview, questionnaires, actigraphy, and sleep log data as well as meeting other eligibility criteria.
  Interventions: Behavioral: Serial awakenings
- Healthy sleeping controls: Participants classified as having healthy sleepy through clinical interview, questionnaires, actigraphy, and sleep log data as well as meeting other eligibility criteria.
  Interventions: Behavioral: Serial awakenings

INTERVENTIONS:
Behavioral: Serial awakenings — The first study night will be a baseline sleep recording. The second night will consist of a series of awakenings (using auditory tones) and subsequent periods of falling back asleep in order to examine the cortical dynamics of hyperarousal or other dysfunction during these two critical sleep processes in insomnia.

SUMMARY:
Insomnia, defined as a subjective report of difficulty initiating sleep, maintaining sleep, and/or non-restorative sleep, leads to significant daytime dysfunction and increased health risks. A commonly held hypothesis is that insomnia is caused by a state of hyperarousal, but the neurobiological mechanisms of hyperarousal in insomnia are poorly understood, in part because of limitations in our ability to image the brain during normal human sleep with sufficient temporal resolution. Furthermore, the efficacy of insomnia treatment is judged by subjective report of the patient and demonstration of changes in sleep latency and/or sleep amount which are generally small in magnitude; there are currently no data to demonstrate that insomnia treatments correct any functional abnormalities in the sleep process that likely contribute to neurobehavioral abnormalities and health risks. The goals of the proposed study are to use high density EEG to define abnormalities in specific aspects of sleep in insomnia patients compared to healthy sleeping control subjects to define biomarkers that will both increase our understanding of the pathophysiology of insomnia as well as provide targets to assess treatments for insomnia.

DETAILED DESCRIPTION:
Recent advances in electroencephalographic recording techniques have produced new ways to probe the process and function of sleep. Through the use of high-density EEG (hdEEG, up to 256 channels), it is possible to approach the spatial resolution of other brain imaging modalities while affording the millisecond temporal resolution of EEG and providing a direct measure of the underlying brain activity, unlike the indirect and/or secondary biophysical signals of brain hemodynamics/metabolism obtained with PET or SPECT that are suboptimal for exploring the short-lived spatio-temporal dynamics of many brain processes.

Here we used hdEEG to try to characterize topographic changes in sleep EEG expression in individuals with insomnia compared to normal controls. We further used serial awakenings to determine if individuals with insomnia were more likely to subjectively report being awake when they were sleeping, and study instances where a direct confirmation of sleep was followed by a subjective report of wakefulness to see if they are characterized by changes in EEG oscillations.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* English speaking, reading, and writing
* For control subjects: Insomnia Severity Index (ISI) less than or equal to 6 and does not meet criteria for insomnia
* For insomnia subjects: ISI greater than or equal to 7, meets criteria for insomnia, and reports insomnia symptoms for at least 6 months

Exclusion Criteria:

* Imminent danger to self or others
* Clinical diagnosis of dementia
* Active Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV Axis I disorder or alcohol or drug dependence or abuse
* Other sleep disorders aside from insomnia
* History of significant head trauma or loss of consciousness over 30 minutes
* Regular use of psychotropic medications in past 4 weeks
* Regular tobacco use
* Drinking more than 3 caffeinated beverages per day
* Significant neurological or medical illness
* Pregnant, less than 6 months post-partum, or planning to become pregnant during the study
* Left-handedness
* Body Mass Index (BMI) greater than 40
* Apnea Hypopnea Index (AHI) greater than 10 on Apnea Link
* Mini mental status exam score less than 27

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the community and from patients presenting at the Wisconsin Sleep and UW-Psychiatry clinics for insomnia.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith E Rumble, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Sleeping Controls: Participants classified as having healthy sleep through clinical interview, questionnaires, actigraphy, and sleep log data as well as meeting other eligibility criteria.
Period: Overall Study
Arm/Group | Primary Insomnia | Healthy Sleeping Controls
Started | 23 | 22
Completed | 17 | 17
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Sleep apnea in Night 1 | 1 | 0
Not completed — Poor Sleep in Night 1 | 0 | 2
Not completed — No Sex/Age Match Night 1 | 1 | 0
Not completed — No Sex/Age Match Night 2 | 0 | 2
Not completed — Technical Difficulties Night 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Insomnia | Healthy Sleeping Controls | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (8.2) | 31.1 (8.1) | 30.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) is a questionnaire that assesses insomnia severity over the course of the previous 2 weeks and provides evidence for our study groups. The ISI includes seven items, which measure insomnia symptom severity on a five-point scale ranging from 0 (not at all) to 4 (very much). The ISI score is obtained by adding individual item scores (possible range of 0-28), with higher scores indicating greater insomnia severity.
  units on a scale | 14.8 (3.1) | 1.2 (1.5) | 8.0 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: EEG Power During Sleep
Description: The difference in spontaneous NREM sleep (stage N2 or N3) EEG power between subjects with insomnia and good sleeping controls measured with 256 channel high-density EEG equipment. Reported here is the median spectral power estimated using Welch's method (MATLAB function pwelch) across all 6 second epochs staged by a registered sleep technician as NREM sleep stage N2 or N3 sleep. The median spectral estimate across all NREM epochs was used to estimate spectral power for each subject as this value is robust to outliers from individual sleep epochs. The Welch's method done in this way estimates frequency content in .33 Hz bins which are then averaged across the spindle frequency band range (12 - 16Hz) from the approximate CP1 electrode (channel 89). The value reported below is the MEAN of the median spectral estimate. Higher values represent more spindle band activity. This frequency range and location showed the most consistent difference between groups across outcome measures.
Time Frame: Individual night of sleep recorded on average within 4 weeks of enrollment (Night 1, Baseline EEG)
Measure: Mean (Full Range); unit: μV^2/Hz
Groups:
- Primary Insomnia: An initial baseline 256 channel high-density EEG polysomnographic recording was acquired using an Electrical Geodesics NetAmps 300 System (256 EEG channels) integrated with clinical polysomnography (PSG) from the Alice 5 Sleepware system (hdPSG). This baseline recording included electrooculogram (EOG), chin and leg electromyography (EMG), electrocardiogram (EKG), blood oxygen level (SpO2), respiration belts, a snore microphone and a position sensor and was used to rule out clinical sleep disorders other than insomnia. Lights off typically occurred within 30 minutes of subjects normal sleep time and subjects were allowed to sleep ad libitum. Sleep staging and arousal detection was performed by a sleep technician according to American Academy of Sleep Medicine standard criteria. Data was included for all subjects who completed the sleep recording and had a suitable sex and age matched control.
- Healthy Sleeping Controls: An initial baseline 256 channel high-density EEG polysomnographic recording was acquired using an Electrical Geodesics NetAmps 300 System (256 EEG channels) integrated with clinical polysomnography (PSG) from the Alice 5 Sleepware system (hdPSG). This baseline recording included electrooculogram (EOG), chin and leg electromyography (EMG), electrocardiogram (EKG), blood oxygen level (SpO2), respiration belts, a snore microphone and a position sensor and was used to rule out clinical sleep disorders. Lights off typically occurred within 30 minutes of subjects normal sleep time and subjects were allowed to sleep ad libitum. Sleep staging and arousal detection was performed by a sleep technician according to American Academy of Sleep Medicine standard criteria. Data was included for all subjects who completed the sleep recording and had a suitable sex and age matched insomnia participant.
Arm/Group | Primary Insomnia | Healthy Sleeping Controls
Number analyzed (Participants) | 19 | 19
μV^2/Hz | 1.40 [0.68 to 3.17] | 1.17 [0.38 to 2.46]
Statistical Analysis 1: Comparison: Primary Insomnia vs Healthy Sleeping Controls; Only reporting values for approximate 10-20 channel CP1; Test type: Other — Group comparison, for absolute (spatially z-score normalized across all electrodes for each subject); p = 0.2791, t-test, 2 sided
Statistical Analysis 2: Comparison: Primary Insomnia vs Healthy Sleeping Controls; Test type: Other — Group comparison, for absolute multiple comparisons correction across electrodes using threshold free cluster enhancement (TFCE); p = 0.9, t-test, 2 sided

2. Primary Outcome: EEG Power Examined Before Arousal From Sleep on Serial Awakening Night
Description: The difference in 30 seconds of spontaneous NREM (stage N2 or N3) sleep EEG power prior to serial awakening between subjects with insomnia and good sleeping controls measured with 256 channel high-density EEG equipment. Reported here is the median spectral power estimated using Welch's method (2 second epochs) of the 30 seconds of NREM sleep stage N2 or N3 sleep immediately prior to the 40dB tone played to initiate a serial awakening sequence. The median spectral estimate across epochs was used to estimate spectral power for each subject as this value is robust to outliers from individual epochs. The Welch's method done in this way estimates frequency content in .5 Hz bins which are then averaged across the spindle frequency band range (12 - 16Hz) from the approximate CP1 electrode (channel 89). Each subject had between 4 - 10 serial awakenings from NREM sleep. The value reported below is the MEAN of the median spectral estimate. Higher values represent more spindle band activity.
Time Frame: 30 seconds of NREM sleep prior to serial awakening (Night 2, Serial Awakening EEG)
Measure: Mean (Full Range); unit: μV^2/Hz
Groups:
- Primary Insomnia; Healthy Sleeping Controls: After the baseline sleep night participants returned to the sleep lab the following night for the serial awakening night. During the day they were asked to follow their usual schedule of activities and were instructed not to nap. Returning participants were outfitted with the hdEEG net in addition to EOG, chin EMG and EKG leads, along with small, comfortable sleep specific headband speakers (SleepPhones) covering the ears, through which the experimenter could talk to the subject and computer-generated sounds could be played. The headband speakers were secured with gauze to prevent movement during the night. After the onset of stable sleep, participants were probed repeatedly using 10 sec tones (2000 hertz (Hz) pure tones) starting at 40 decibels (dB) and increasing by 5 dB every 30 sec until full awakening. Participants were then encouraged to fall back asleep naturally and were only awakened again once they reached stable sleep. No awakenings were attempted after the subject's normal waking time and subjects could sleep ad libitum. Sleep staging and arousal detection was performed in real-time but was also verified offline by a sleep technician blind to the presence of the auditory tone sequence according to American Academy of Sleep Medicine standard criteria. Data from 2 insomnia subjects and their age and sex matched controls was excluded because of technical difficulties with the hdEEG recording.
Arm/Group | Primary Insomnia | Healthy Sleeping Controls
Number analyzed (Participants) | 17 | 17
μV^2/Hz | 1.20 [0.59 to 2.09] | 0.93 [0.22 to 1.70]
Statistical Analysis 1: Comparison: Primary Insomnia vs Healthy Sleeping Controls; Only reporting values for approximate 10-20 channel CP1; Test type: Other — Group comparison, for both absolute (spatially z-score normalized across all electrodes for each subject); p = 0.1069, t-test, 2 sided
Statistical Analysis 2: Comparison: Primary Insomnia vs Healthy Sleeping Controls; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.546, t-test, 2 sided

3. Primary Outcome: EEG Power Examined as Subjects Fall Asleep on Serial Awakening Night
Description: The difference in 30 seconds of spontaneous falling asleep EEG power between subjects with insomnia and good sleeping controls measured with 256 channel high-density EEG equipment. Reported here is the median spectral power estimated using Welch's method with 2 second epochs from the 30 seconds of sleep immediately following a serial awakening (starting after the last waking epoch) that resulted in the subject reaching 5 minutes of stable sleep averaged across the spindle frequency band range 12 - 16Hz from the approximate CP1 electrode (channel 89) and across all serial awakening falling asleep periods for each subject. Each subject had between 4 - 8 falling asleep periods that resulted in 5 minutes of stable sleep within 30 minutes of the serial awakening attempt. The value reported below is the MEAN of the median spectral estimate. Higher values represent more spindle band activity.
Time Frame: 30 seconds of falling asleep EEG immediately after the first non-waking epoch following a serial awakening and proceeding 5 minutes of stable sleep (Night 2, Serial Awakening EEG)
Measure: Mean (Full Range); unit: μV^2/Hz
Arm/Group | Primary Insomnia | Healthy Sleeping Controls
Number analyzed (Participants) | 17 | 17
μV^2/Hz | 0.57 [0.42 to 2.09] | 0.50 [0.39 to 1.00]
Statistical Analysis 1: Comparison: Primary Insomnia vs Healthy Sleeping Controls; Only reporting values for approximate 10-20 channel CP1; Test type: Other — Group comparison, for absolute (spatially z-score normalized across all electrodes for each subject); p = 0.2918, t-test, 2 sided
Statistical Analysis 2: Comparison: Primary Insomnia vs Healthy Sleeping Controls; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.761, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at all study visits, including overnight visits, over ~4 weeks of participation.
Arm/Group | Primary Insomnia | Healthy Sleeping Controls
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT01960452/Prot_SAP_000.pdf